CLINICAL TRIAL: NCT01380366
Title: Influence of Recombinant Human Growth Hormone on Intestinal Permeability and Liver Injury in Intestinal Failure Patients Receiving Parenteral Nutrition (Serono Project)
Brief Title: rHGH and Intestinal Permeability in Intestinal Failure
Acronym: rHGH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Northwestern Memorial Hospital (Other); EMD Serono (Industry)
Responsible Party: Principal Investigator, Jonathan Fryer, Associate Professor in Surgery-Organ Transplantation, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00012123 0208-007; CNV0050754 (Other: Internal Tracking Sponsor Contract ID)
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Short Bowel Syndrome
Keywords: Malabsorption
MeSH Terms: conditions — Short Bowel Syndrome; Malabsorption Syndromes | interventions — Human Growth Hormone; Growth Hormone; Diet Records; Hematologic Tests; Standard of Care; Angptl4 protein, mouse; Urine Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients consent to rHGH study (Other): Patients consent to be given growth hormone (rHGH) for their short bowel syndrome.
  Interventions: Drug: Somatropin; Procedure: Seven Day Food Diary; Procedure: Blood Tests (standard of care); Other: Fasting; Other: Sugar Permeability Test; Other: Urine Collection

INTERVENTIONS:
Drug: Somatropin — Patients are given somatropin (growth hormone) for their short bowel syndrome for 28 days at a dose of 0.1 mg/kg subcutaneously daily to a maximum of 8 mg daily.
  Other Names: Recombinant human growth hormone (rHGH); Zorbtive®
Procedure: Seven Day Food Diary — Subjects are asked to fill out a seven day food diary the week prior to their inpatient appointment, prior to receiving rHGH treatment for their short bowel syndrome. Subjects will be asked to repeat the use of a food diary after completing the administration of the growth hormone.
Procedure: Blood Tests (standard of care) — Blood tests are taken (standard of care) to evaluate the potential hepato-protective effects of improving intestinal barrier function on those receiving human growth hormone for short bowel syndrome. Per clinical protocol to test liver function i.e. Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline phosphatase (ALP), Gamma-glutamyl transpeptidase (GGT), Total Bilirubin). A complete blood count (CBC) with platelets (PLTS) and white-count differential (WBC with diff) is performed to check for anemia and infection. These tests will be taken at baseline (before fasting) and repeated again on the 28th day (last dose) of the growth hormone. Blood is also taken at clinical visit over the next two years (approximately every two months).
Other: Fasting — Eight hour overnight fast prior to being given sucralose, mannitol, lactulose, and sucrose. This is done at baseline (day one) and repeated again after the last dose of growth hormone and prior to sugar permeability urine tests.
Other: Sugar Permeability Test — Subject will be given 4 capsules of sucralose (250mg per capsule), 2.0 grams of mannitol, 7.5 grams of lactulose, and 40 grams of sucrose in 150 mL of water. This will be given on the second day of the study after an 8-hour overnight fast and repeated within 72 hours of the last dose of growth hormone.
Other: Urine Collection — Urine will be collected for the following five hours after subject has been given combination of sucralose, mannitol, lactulose, and sucrose to complete the intestinal sugar permeability test looking at urine ratio of lactulose to mannitol (L/M ratio). Tests include urinalysis (UA) and a blood urea nitrogen (BUN)/creatinine (Cr).

SUMMARY:
Patients who are being asked to participate in this study have a short small bowel and will be prescribed to take the medication: Zorbtive® ("Zorbtive/Somatropin/(rHGH)"). Zorbtive® is an FDA approved recombinant human growth hormone (rHGH). The investigators want to see if taking this medication improves small bowel function by helping it to take in food, nutrients, vitamins and minerals. The investigators also believe that if the small bowel is absorbing food and nutrients better, liver function will improve as well. Therefore, liver function will also be monitored during the course of the study by performing blood tests.

DETAILED DESCRIPTION:
This is an open-label pilot study in which a convenience sample of 20 subjects will participate for up to 26 months.

At the baseline visit, subjects will sign a consent form after all questions they have are answered. An inpatient appointment will be made at the General Clinical Research Center (GCRC). Subjects will be given instructions to fill out a 7-day food diary the week prior to their inpatient appointment. In this diary, subjects will be asked to record the types and amounts of food they ingest over a 7-day period. This will allow researchers to review subjects' food intake prior to sugar permeability testing. Although each subject serves as his/her own control, this information may be useful upon review of variations in permeability between subjects.

To evaluate the potential hepato-protective effects of improving intestinal barrier function, blood tests evaluating liver injury and function (i.e. ALT, AST, total bilirubin, ALP, GGT) will be obtained. These labs are part of the subject's standard of care follow-up, therefore study staff will abstract these data from the subject's medical record. The sugar permeability testing requires an 8-hour overnight fast, followed by the ingestion of 4 capsules of sucralose (250mg per capsule), 2.0 grams of mannitol, 7.5 grams of lactulose, and 40 grams of sucrose in 150 mL of water. Over the next 5 hours, urine is collected. Intestinal permeability is quantified as the urine ratio of lactulose, mannitol and sucralose. After urine collection is complete, subjects will begin their 28 days of Zorbtive® administration.

All evaluations (subject food diary, bloodwork, and sugar permeability testing) will be repeated 28 days later, within 72 hours of receiving the final dose of Zorbtive®. The bloodwork drawn is part of the subject's standard of care follow-up, therefore study staff will abstract these data from the subject's medical record.

Following completion of study visits at the GCRC, study staff will obtain results of liver injury/ function tests [(ALT), (AST), bilirubin, alkaline phosphatase (ALK or ALP), (GGT)] from the medical record from each routine clinical exam from Month 3 through Month 24, following the 28-day treatment with Zorbtive® therapy. These labs are part of the subject's standard of care follow-up, therefore study staff will abstract these data from the subject's medical record. Subjects will not be asked to return for separate study visits.

Since the intestinal epithelium is completely reconstituted approximately every 7 days, it is anticipated that the potential influences of rHGH on barrier function and related liver injury will be realized by the end of the 28 day study period. The long term durability of any changes observed after 28 days will be observed, but will likely require further study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between the ages of 18 and 80
* Subjects can be male or female
* Subjects must have short bowel syndrome with <200cm of functional small bowel or have severe small bowel dysfunction mandating regular (at least two times per week) administration of total parenteral nutrition (TPN) and/or IV fluids.
* Subjects must have been dependent on TPN or IV fluids for 1 year, or are expected to be dependent on TPN or IV fluids for at least 1 yr.
* Subjects must be patients being seen in the Northwestern intestinal failure clinic
* Subjects must be willing to spend one night in the Clinical Research Center
* Subjects must be able to read, understand and be able to sign the study specific informed consent

Exclusion Criteria:

* Subjects must be greater than or equal to 18 years of age, but less than or equal to 80 years of age
* Infections requiring antibiotic therapy within one week of starting the study
* Subjects must not have evidence of an ongoing malignancy for two years
* Subjects must not have history of antibiotic use within one week of initiating the study. Subjects may enroll in the study as long as Visit 1 is at least one week from the last dose of antibiotics.
* Subjects that have evidence of acute critical illness due to complications following open heart or abdominal surgery, multiple accidental trauma, or acute respiratory failure
* Subjects with known liver disease, positive hepatitis B virus (HBV), or hepatitis C virus (HCV) serology
* Subjects unwilling to abstain from alcohol 7 days prior to and during the 28 days of Zorbtive® therapy, until completion of Visit 2
* Subjects with a known sensitivity to Benzyl Alcohol
* Subjects with a known sensitivity to growth hormone
* Female subjects that are unable or unwilling to use effective, acceptable birth control methods throughout the study and for up to 6 months after completing treatment with Zorbtive therapy
* Female subject with a positive pregnancy test

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-10; Primary Completion 2011-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Fryer, MD, Principal Investigator — Northwestern Memorial Hospital, Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Zorptive Subjects: Patients consent to rHGH and Intestinal Permeability in Intestinal Failure Study
Period: Overall Study
Arm/Group | Zorptive Subjects
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients Consented to be Given rHGH
Groups:
- Patients Consented to be Given rHGH: Patients given growth hormone (rHGH) for their short bowel syndrome.
Arm/Group | Patients Consented to be Given rHGH
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (15.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: To Identify Small Intestinal Permeability Changes in Short Bowel Syndrome Patients After Administration of Recombinant Human Growth Hormone (Zorbtive®).
Description: Permeability changes will be identified in short bowel syndrome patients by evaluating concentration of lactulose, mannitol and sucralose from Visit 1 to Visit 2. A decrease in concentration of sucralose in urine indicates Zorbtive potentially enhancing intestinal barrier function.
Time Frame: (Visit 1) Baseline to (Visit 2) 28-31 days after baseline
Measure: Number; unit: participants
Groups:
- Patients Experiencing Decrease in Concentration of Sucralose: A decrease in concentration of sucralose in urine indicates Zorbtive potentially enhancing intestinal barrier function.
Arm/Group | Patients Experiencing Decrease in Concentration of Sucralose
Number analyzed (Participants) | 7
participants | 7

2. Secondary Outcome: To Evaluate Liver Enzymes in Total Parenteral Nutrition (TPN)-Dependent Short Bowel Syndrome Patients Before and After Administration of Zorbtive®.
Description: Following completion of Visit 2, study staff will obtain results of liver injury/function tests (ALT, Aspartate transaminase (AST), bilirubin, alkaline phosphatase (ALK or ALP), GGT) from the medical record from each routine clinical exam from Month 3 through Month 24. Results that show decreased liver injury (ALT, AST, bilirubin, alkaline phosphate (ALK or ALP), GGT) will show Zorbtive administration enhanced intestinal permeability and enhanced liver function.
Time Frame: (Visit 1) Baseline, (Visit 2) 28-31 days after baseline, then at regularly scheduled follow-up clinic visits for two years from Month 3 through Month 24
Measure: Number; unit: participants
Groups:
- Patient Decreased Liver Injury: Results that show decreased liver injury (ALT, AST, bilirubin, alkaline phosphate (ALK or ALP), GGT) will show Zorbtive administration enhanced intestinal permeability and enhanced liver function.
Arm/Group | Patient Decreased Liver Injury
Number analyzed (Participants) | 7
participants | 7

ADVERSE EVENTS:
Time Frame: Up to 2 years after enrollment.
Arm/Group | Patients Consented to be Given rHGH
Serious Adverse Events (participants affected / at risk) | 6/15
Other Adverse Events (participants affected / at risk) | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Consented to be Given rHGH (N=15)
Hospitalization for Escherichia coli Infection (Blood and lymphatic system disorders) | 1 (1)
Hospitalization for Gram-positive Cocci (Blood and lymphatic system disorders) | 1 (1)
Hospitalization for positive line infection (Blood and lymphatic system disorders) | 1 (1)
Pancreatitis (Endocrine disorders) | 1 (1)
Hospitalization for abdominal pain (pre-treatment) (Gastrointestinal disorders) | 1 (1)
Hospitalization for Flu like Symptoms (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
Number of participants is low. Time period of evaluation may not have been adequate for evaluating the impact on liver injury. Parameters used to evaluate the impact of gut permeability changes on hepatic inflammation and injury were very limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes